CLINICAL TRIAL: NCT06782139
Title: Effects of ENavogliflozin on Coronary microVascular and Cardiac Function in Patients With obesitY (ENVY)
Brief Title: Effects of Enavogliflozin on Coronary Microvascular and Cardiac Function in Obesity
Acronym: ENVY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Seong-Mi Park, M.D. Ph.D., Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024AN0301
Record Dates: First submitted 2024-12-09; First posted 2025-01-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Obesity and Type 2 Diabetes
Keywords: Sodium-Glucose Cotransporter 2 inhibitors; Obesity; Diabetes; Coronary microvascular function; Epicardial adipose tissue
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enavogliflozin (Experimental): The medication is a soft, orange, bi-convex, triangular film-coated tablet, and it is administered once daily at a dose of 0.3 mg, regardless of meals.
  Interventions: Drug: Enavogliflozin
- Placebo (Placebo Comparator): The placebo is provided by the pharmaceutical company in the form of a tablet that is identical in size, shape, taste, and odor to the active intervention medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enavogliflozin — Patients who are enrolled in the study will undergo adenosine stress tests assessing coronary flow velocity reserve and body composition analysis on the day of registration. Within 2 weeks, cardiopulmonary exercise tests will be performed with exhalation gas analysis. After completing the baseline cardiopulmonary exercise capacity evaluation, patients will be assigned to either the enavogliflozin or placebo group and monitored for adverse effects within one month. Patients without significant adverse effects will continue the assigned treatment, and at 12 weeks, they will undergo re-evaluation of coronary flow velocity reserve, body composition analysis, and cardiopulmonary exercise capacity. Adverse events will be monitored from the date of enrollment through the final evaluation.
  Arms: Enavogliflozin
Drug: Placebo — Patients who are enrolled in the study will undergo adenosine stress tests assessing coronary flow velocity reserve and body composition analysis on the day of registration. Within 2 weeks, cardiopulmonary exercise tests will be performed with exhalation gas analysis. After completing the baseline cardiopulmonary exercise capacity evaluation, patients will be assigned to either the enavogliflozin or placebo group and monitored for adverse effects within one month. Patients without significant adverse effects will continue the assigned treatment, and at 12 weeks, they will undergo re-evaluation of coronary flow velocity reserve, body composition analysis, and cardiopulmonary exercise capacity. Adverse events will be monitored from the date of enrollment through the final evaluation.
  Arms: Placebo

SUMMARY:
The goal of this study is to analyze the effects of enavogliflozin on heart function and coronary microvascular function in obese patients compared to a placebo, and to evaluate the improvement in cardiopulmonary exercise capacity in these patients.

DETAILED DESCRIPTION:
In recent years, the prevalence of obesity has increased, which acts as a significant risk factor for cardiovascular diseases. Obesity is closely related to reduced microvascular function, increased insulin resistance, and elevated blood pressure, and it is particularly known to be a major cause of heart failure with preserved ejection fraction (HFpEF) and diastolic dysfunction. Coronary microvascular dysfunction (CMD) leads to angina, myocardial infarction, and heart failure, which are associated with increased mortality. CMD has recently gained more importance as one of the key mechanisms of HFpEF. However, CMD often shows poor response to standard treatments, and when not recognized by healthcare providers, it can result in poor outcomes due to a lack of appropriate treatment.

Sodium-Glucose Cotransporter 2 (SGLT2) inhibitors are drugs that inhibit glucose reabsorption by blocking SGLT2 in the proximal tubules of the kidneys, thereby lowering blood sugar. Initially developed as oral hypoglycemic agents, previous randomized controlled studies have shown that they also have significant beneficial effects on heart failure and cardiovascular diseases not only in diabetic patients but also in non-diabetic patients. Recent studies have also demonstrated the effectiveness of SGLT2 inhibitors in patients with HFpEF. SGLT2 inhibitors reduce excessive sodium excretion through urine, which reduces fluid volume, lowers blood pressure, and decreases body weight, but the exact mechanism of their significant effects in cardiovascular diseases is still not fully understood. In particular, research on the effects of SGLT2 inhibitors on microvascular function is still limited. Recently, a randomized controlled study involving 16 diabetic patients reported an increase in myocardial flow reserve after 4 weeks of dapagliflozin administration, while another study involving 90 high-risk cardiovascular diabetic patients showed no significant change in myocardial flow reserve at 13 weeks with empagliflozin. Regarding enavogliflozin, a recent animal study in pigs suggested that it could improve vascular function by intervening in coronary endothelial cell function.

This study hypothesized that enavogliflozin would improve microvascular abnormalities and enhance heart function and cardiopulmonary exercise capacity in obesity-related cardiovascular diseases. Therefore, the objective of this study is to analyze the effects of enavogliflozin on heart function and microvascular function in obese patients compared to a placebo, and to evaluate the improvement in cardiopulmonary exercise capacity in these patients.

ELIGIBILITY:
Inclusion Criteria: The following criteria must be met for inclusion in the study:

1. Obesity or Abdominal Obesity:

   Body Mass Index (BMI) ≥ 25 kg/m², or Waist circumference: Male ≥ 90 cm, Female ≥ 85 cm.
2. Diabetes:

Hemoglobin A1c ≥ 6.5%, or Fasting blood glucose ≥ 126 mg/dL after 8 hours of fasting, or Currently on antidiabetic medication. Blood test results must be within 3 months prior to enrollment.

Other inclusion criteria:

Age between 20 and 79 years. Patients who have undergone coronary flow velocity reserve testing. For baseline echocardiography, left ventricular diastolic dysfunction will be evaluated structurally (LV dimension, LV mass index, LA size) and hemodynamically (Doppler data, left ventricular ejection fraction, strain data).

Exclusion Criteria:

1. Left ventricular ejection fraction (LVEF) < 50%
2. History of coronary artery disease, or patients who have undergone coronary artery intervention or coronary artery bypass grafting.
3. Patients with suspected obstructive coronary artery disease, including those with chest pain and positive stress test results (e.g., exercise treadmill test, dobutamine stress echocardiography, myocardial perfusion imaging).
4. Second-degree or higher atrioventricular block, symptomatic bradycardia, sick sinus syndrome, or Wolff-Parkinson-White syndrome.
5. Chronic kidney disease (GFR < 30 mL/min/1.73 m²) or end-stage renal disease on hemodialysis or peritoneal dialysis.
6. Asthma, chronic obstructive pulmonary disease, or primary pulmonary hypertension.
7. Moderate or severe valvular heart disease or congenital heart disease, or patients with a history of open-heart surgery.
8. Active cancer within the last 5 years, or patients currently receiving chemotherapy.
9. Vasculitis associated with autoimmune diseases, such as systemic lupus erythematosus (SLE) or rheumatoid arthritis (RA).
10. Patients who cannot undergo exercise testing, such as treadmill or bicycle ergometer testing.
11. Use of any other SGLT2 inhibitors (e.g., dapagliflozin, empagliflozin) within the past 6 months, or a known allergy to these drugs.
12. Pregnant or breastfeeding women.
13. Women planning pregnancy during the study period (or within 24 weeks from the start of the study, including the 12-week observation period).
14. Acute urinary tract infection at the time of enrollment.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary microvascular function | From enrollment to the end of treatment at 12 weeks
  The changes in coronary flow velocity reserve at 12 weeks compared to baseline in the active drug/placebo groups

SECONDARY OUTCOMES:
Cardiopulmonary exercise capacity (VO2peak, mL/min/kg) | From enrollment to the end of treatment at 12 weeks
  The changes in cardiopulmonary exercise capacity ((VO2peak, mL/min/kg) at 12 weeks compared to baseline in the active drug/placebo groups
Body weight (kg) | From enrollment to the end of treatment at 12 weeks
  Changes in body weight (kg) at 12 weeks compared to baseline
Systolic and diastolic blood pressure (mmHg) | From enrollment to the end of treatment at 12 weeks
  Changes in Systolic and diastolic blood pressure (mmHg) at 12 weeks compared to baseline
Waist circumference (cm) | From enrollment to the end of treatment at 12 weeks
  Changes in waist circumference (cm) at 12 weeks compared to baseline
Lipid profile | From enrollment to the end of treatment at 12 weeks
  Changes in total cholesterol (mg/dL), triglycerides (mg/dL), high-density lipoprotein cholesterol (mg/dL), and low-density lipoprotein cholesterol (mg/dL) at 12 weeks compared to baseline
Hemoglobin A1c (%) | From enrollment to the end of treatment at 12 weeks
  Changes in hemoglobin A1c (%) at 12 weeks compared to baseline
NT-proBNP (pg/mL) | From enrollment to the end of treatment at 12 weeks
  Changes in NT-proBNP (pg/mL) at 12 weeks compared to baseline
Self-assessment of sarcopenia (score) | From enrollment to the end of treatment at 12 weeks
  Changes in self-assessment of sarcopenia (score) at 12 weeks compared to baseline
5-time chair rise test (sec) | From enrollment to the end of treatment at 12 weeks
  Changes in 5-time chair rise test (sec) at 12 weeks compared to baseline
Body composition analysis - skeletal muscle mass index | From enrollment to the end of treatment at 12 weeks
  Changes in skeletal muscle mass index (kg/m2) at 12 weeks compared to baseline
Body composition analysis - visceral fat area | From enrollment to the end of treatment at 12 weeks
  Changes in visceral fat area (cm2) at 12 weeks compared to baseline
Echocardiographic findings - chamber size (mm) | From enrollment to the end of treatment at 12 weeks
  Changes in chamber size (mm) at 12 weeks compared to baseline
Echocardiographic findings - ejection fraction (%) | From enrollment to the end of treatment at 12 weeks
  Changes in ejection fraction (%) at 12 weeks compared to baseline
Echocardiographic findings - E/e' | From enrollment to the end of treatment at 12 weeks
  Changes in E/e' at 12 weeks compared to baseline
Echocardiographic findings - global longitudinal strain (%) | From enrollment to the end of treatment at 12 weeks
  Changes in global longitudinal strain (%) at 12 weeks compared to baseline
Epicardial Adipose tissue | % change of EAT from baseline to 12weeks
  % change of EAT from baseline to 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Mi Park, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No